CLINICAL TRIAL: NCT00975039
Title: Evaluation of the Safety and Efficacy of WST11-mediated Vascular Targeted Photodynamic Therapy in Non-resectable or Inoperable Cholangiocarcinoma
Brief Title: Study Using WST11 in Patients With Non-Resectable or Inoperable Cholangiocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early end of enrolment with regards to difficulty met to enrol patients .
Sponsor: Steba Biotech S.A. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLIN904 CCM201
Record Dates: First submitted 2009-09-10; First posted 2009-09-11 (Estimated); Last update posted 2016-04-18 (Estimated); Status verified 2016-04

CONDITIONS: Cholangiocarcinoma
Keywords: Inoperable; Inoperable Cholangiocarcinoma; Non-resectable; Non-resectable Cholangiocarcinoma; Carcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Carcinoma | interventions — padeliporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- WST11 (Experimental): Treatment with WST11-mediated VTP
  Interventions: Drug: WST11

INTERVENTIONS:
Drug: WST11 — WST11-mediated VTP will consist of the combination of a single IV administration of WST11 at doses of 2.5 and 5 mg/kg, using 753nm laser light at a fixed power (150 mW/cm) and light energy (200 J/cm). Illumination in the bile duct is performed by inserting a diffusing fiber, with cylindrical uniform light distribution, in a transparent standard ERCP catheter and by positioning, under radioscopy, the illumination tip of the diffusing fiber in front of the lesion.
  Other Names: WST11-mediated VTP

SUMMARY:
The aim of this study is to evaluate the safety of Vascular Targeted Photodynamic therapy with WST11 in patients with non-resectable or inoperable biliary carcinoma.

DETAILED DESCRIPTION:
This is an open-label, prospective, multicentre, phase IIa study, evaluating a new therapeutic agent in the management of patients suffering from inoperable or non resectable biliary carcinoma. The patients will receive the dose of WST11 according to order of inclusion. The first 3 patients will receive 2.5 mg/kg. In the absence of toxicity, the following 9 patients will receive the dose of 5 mg/kg.

The patient is to receive anesthesia. WST11-mediated therapy will consist of the combination of single IV administration of WST11 at doses of 2.5mg/kg or 5mg/kg, using 753nm laser light at a fixed power of (150mW/cm) and light energy (200 J/cm) delivered through a diffusing fiber. The fiber is introduced in a transparent standard ERCP catheter and positioned under radioscopy in front of the lesion.

ELIGIBILITY:
Inclusion Criteria:

* Patient having signed the consent form to take part in the study
* Patient aged over 18 years, with no upper age limit
* Patient with histologically proven cholangiocarcinoma
* Patient with cholangiocarcinoma, inoperable or non resectable owing to extension, age or concomitant diseases
* Bilirubin level decrease of more than 50% after stent insertion compared to base level
* Patient with a WHO Performance Scale ≤ 2
* Patient in whom efficient drainage is performed by means of a plastic biliary stent endoscopically or radiologically
* Patient capable of completing the quality of life questionnaires
* Women of child-bearing potential must have a negative pregnancy test, and must thereafter prove to be using acceptable contraception (oral contraceptive pill, hormone patches, or IUD)

Exclusion Criteria:

* Absence of consent to take part in the study
* Patient with operable biliary carcinoma
* Class ASA IV patients
* Patients presenting clinical and laboratory signs of biliary infection
* Absence of bilirubin decrease after stent insertion
* Patients with extrinsic biliary compression
* Patients already having received or currently receiving radiotherapy or chemotherapy for cholangiocarcinoma or needing to be treated during the first month of the follow-up
* Known metastatic lesions
* Patients having received immediate treatment by insertion of a metal stent
* Patients with porphyria or known hypersensitivity to porphyrins (contraindication to WST11)
* Patient receiving prohibited treatment at the time of inclusion in the study
* Pregnant or breast-feeding women
* Non-menopausal women not using effective contraception
* Majors under protection as per the French Public Health Code
* Persons not registered with or covered by a social security system
* Persons in an exclusion period relative to other biomedical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety based on analysis of adverse events , clinical laboratory tests, electrocardiogram, physical examination, absence of local or general complications and phototoxicity of WST11 in inoperable or non resectable cholangiocarcinoma | Patient inclusion - Month 6

SECONDARY OUTCOMES:
Evaluation of the antitumor efficacy of WST11-mediated VTP therapy by comparing the objective response rate on the tumor. | Month 1, Month 3 & Month 6
Evaluation of the effect of WST11-mediated VTP therapy on cholestasis and on the incidence of biliary complications of obstructive origin. | Month 1, Month 3 & Month 6
Evaluation of the effect of treatment on patient quality of life QLQ-C30. | Month 1, Month 3 & Month 6
Evaluation of the global survival after WST11-mediated VTP | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Ben Soussan, MD, Principal Investigator — Clinique de l'Alma
Locations (1):
- Clinique de l'Alma, Paris, France

IPD SHARING:
Plan to Share IPD: No